CLINICAL TRIAL: NCT01895036
Title: Nalrexone Facilitated Discontinuation of Buprenorphine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elias Dakwar, research psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6332
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Stable Opioid Dependence
Keywords: maintained on 2 mg or less of buprenorphine, in which discontinuation of agonist treatment is clinically feasible but difficult
MeSH Terms: interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Naltrexone (Experimental): PO naltrexone titration on a mixed inpatient/outpatient basis, followed by administration of Vivitrol four days following the 1st dose of naltrexone
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone
  Other Names: Vivitrol

SUMMARY:
The efficacy of buprenorphine as a long-term agonist treatment has been offset by the emergence of intolerable withdrawal phenomena in a subset of individuals on chronic maintenance who attempt to discontinue the medication. Efforts are needed to better understand these challenges encountered with buprenorphine, as well as to develop interventions to facilitate medication discontinuation.

Emerging evidence suggests that these difficulties may be related to the unique effects of buprenorphine on sites other than mu-opioid receptors, such as kappa-opioid receptors. Kappa-opioid agonism produces aversive, dysphoric-like effects, and can also increase the likelihood of reinstatement to drug use through stress-mediated mechanisms. Some of the discomfort observed during drug taper may therefore be due to the attenuation or loss of kappa-opioid antagonism afforded by buprenorphine, as well as to rebound kappa-opioid activation. Naltrexone represents a promising candidate for extending kappa blockade and therefore for facilitating discontinuation attempts. Naltrexone and its active metabolite 6-Beta-naltrexol are competitive antagonists at the mu and kappa receptors, and to a lesser extent at the delta receptor. Naltrexone and buprenorphine have comparable affinity for the mu-opioid receptor and thus buprenorphine is displaced by naltrexone more gradually than are other opioids with less affinity; a careful titration of naltrexone is less likely, therefore, to precipitate severe withdrawal states in individuals coming off buprenorphine, and the two have been combined to good effect in other settings.

The purpose of this study is therefore to investigate the feasibility of naltrexone augmentation on discontinuing buprenorphine in eligible patients on long-term maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, aged 18-49.
2. Currently maintained on buprenorphine, with a clinically acceptable interest in tapering or discontinuing it
3. Willingness to switch over to naltrexone
4. In otherwise good health based on complete medical history, physical examination, vital signs measurement, ECG, and laboratory tests (hematology, blood chemistry, urinalysis) within normal ranges.
5. Able to give informed consent and comply with study procedures,
6. Currently on 2 mg or less of buprenorphine.
7. Voluntarily seeking treatment for opioid dependence.

Exclusion Criteria:

1. Significant current suicidal risk or 1 or more suicide attempts within the past year
2. History of accidental drug overdose in the last three years defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.
3. Positive serum pregnancy test, lactation, or unwillingness to use a satisfactory method of birth control
4. Active psychiatric disorder which might interfere with participation or make participation hazardous, including DSM-IV organic mental disorder, psychotic disorder, or bipolar disorder with mania
5. History of allergic reaction, adverse reaction, or sensitivity to any study medication.
6. Acute hepatitis with SGOT or SGPT > 3 times the upper end of the laboratory normal range (chronic hepatitis is acceptable as we have found naltrexone treatment well tolerate and safe among patients with chronic hepatitis)
7. Currently prescribed or regularly taking opioids for chronic pain
8. Current participation in another intensive psychotherapy or substance abuse treatment program, or participation in another treatment study.
9. Opioid dependence is not well-managed, and characterized by relapses, slips, or missed doses
10. Concurrent treatment with psychotropic medications which may interact adversely with naltrexone, such as duloxetine and valproic acid.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NYSPI, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone: PO naltrexone titration on a mixed inpatient/outpatient basis, followed by administration of Vivitrol four days following the 1st dose of naltrexone
  Naltrexone
Period: Overall Study
Arm/Group | Naltrexone
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Naltrexone
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Successful Discontinuation of Buprenorphine
Description: Number of individuals successfully discontinuing buprenorphine during the inpatient phase and through follow-up.
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: Beginning with entry into the protocol and through 1 month after study completion.
Arm/Group | Naltrexone
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No